CLINICAL TRIAL: NCT01156753
Title: A Phase II, Randomized, Multicenter Study of CDX-011 (CR011-vcMMAE) in Patients With Advanced GPNMB-expressing Breast Cancer
Brief Title: A Study of CDX-011 (CR011-vcMMAE) in Patients With Advanced GPNMB-expressing Breast Cancer
Acronym: EMERGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDX011-03
Record Dates: First submitted 2010-06-30; First posted 2010-07-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: CR011-vcMMAE; locally advanced breast cancer; metastatic breast cancer; breast cancer; CDX-011; GPNMB; Targeted treatment for breast cancer; Locally advanced or metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — glembatumumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CDX-011 (Experimental)
  Interventions: Drug: CDX-011
- "Investigator's Choice" chemotherapy (Active Comparator)
  Interventions: Drug: "Investigator's Choice" chemotherapy

INTERVENTIONS:
Drug: CDX-011 — CDX-011 (1.88 mg/kg) administered as an intravenous infusion on Day 1 of each 21 day cycle.
  Arms: CDX-011
Drug: "Investigator's Choice" chemotherapy — Any of the following single-agent chemotherapy may be given at the discretion of the investigator, with a cycle length not to exceed four weeks: Capecitabine, Vinorelbine, Gemcitabine, Docetaxel, Paclitaxel, Albumin-bound paclitaxel, Doxorubicin HCL, Liposomal doxorubicin, Ixabepilone and Eribulin.
  Arms: "Investigator's Choice" chemotherapy

SUMMARY:
The main purpose of this study is to see whether CDX-011 is effective in treating patients who have advanced breast cancer that makes a protein called glycoprotein NMB (GPNMB), and who have already received (or were not candidates for) all available approved therapies for their breast cancer. This study will also further characterize the safety of CDX-011 treatment in this patient population.

DETAILED DESCRIPTION:
CDX-011 consists of an antibody attached to a drug, monomethyl auristatin E (MMAE), that can kill cancer cells. The antibody delivers the drug to cancer cells by attaching to a protein called glycoprotein NMB (GPNMB) that is expressed on the cancer cell. The MMAE is then released inside of the cell, where it interferes with cell growth and may lead to cell death.

This study will examine the effectiveness and safety of CDX-011 in patients with advanced breast cancer that makes the GPNMB protein. To better assess this, the effect of CDX-011 will be compared to treatment with currently available cancer chemotherapy.

Eligible patients who enroll in the study will be randomly assigned by chance to receive treatment with CDX-011 or with a chemotherapy chosen by their study doctor from a list of currently available drugs ("Investigator's Choice" chemotherapy). For each three patients enrolled, two will receive CDX-011 and one will receive treatment with "Investigator's Choice". Patients initially assigned to "Investigator's Choice" chemotherapy may be offered treatment with CDX-011 if their cancer worsens during this initial treatment.

All patients enrolled in the study will be closely monitored to determine if their cancer is responding to treatment, and for any side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

Among other criteria, patients must meet all of the following conditions to be eligible for the study:

1. 18 years of age or older.
2. Locally advanced or metastatic breast cancer.
3. Previous treatment with at least two but no more than seven prior chemotherapy treatments for progressive, recurrent or metastatic breast cancer.
4. Unless not a candidate for these agents, prior therapies must have included a taxane, an anthracycline, and capecitabine, as well as trastuzumab and lapatinib for patients whose tumors are positive for the human epidermal growth factor receptor 2 (HER2). (Patients who received incomplete courses of therapy with these agents due to intolerance will be eligible.)
5. Breast cancer tumor confirmed to express GPNMB. This will be determined by submitting a tissue sample (obtained during a diagnostic biopsy or surgery) to a central laboratory for analysis.

Exclusion Criteria:

Among other criteria, patients who meet any of the following conditions are NOT eligible for the study:

1. Ongoing neuropathy or other chemotherapy or radiation-related toxicities that are moderate (Grade 2) or worse in severity.
2. Known brain metastases, unless previously treated and asymptomatic for 2 months and not progressive in size or number for 2 months.
3. Significant cardiovascular disease or any other underlying medical condition that, in the Investigator's opinion, will make the administration of study treatment (CDX-011 or chemotherapy) hazardous or would obscure the interpretation of side effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 6 or more weeks following treatment initiation
  The objective response rate (ORR) is defined as the proportion of patients who achieve radiographic partial or complete response (PR or CR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guideline.

SECONDARY OUTCOMES:
Progression-free survival | At least 18 months following treatment initiation
  Progression-free survival is defined as the time from randomization to the earlier of disease progression or death due to any cause.
Adverse Events | Usually following at least 1 cycle of study treatment (1 dose of CDX-011 or "Investigator's Choice" chemotherapy and 3 to 4 weeks of follow-up)
  The number and percentage of patients experiencing one or more adverse events will be summarized by treatment arm, relationship to study drug, and severity.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - The University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Breastlink Medical Group, Long Beach, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Florida Cancer Specialists, West Coast, Florida
  - Peachtree Hematology-Oncology Consultants PC, Atlanta, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Cancer Treatment Centers of America at Midwestern Regional Medical Center, Zion, Illinois
  - Cancer Care of Louisiana, New Orleans, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - Montana Cancer Institute Foundation, Missoula, Montana
  - Clinical Research Alliance Inc., Lake Success, New York
  - Weill Cornell Breast Center/Weill Cornell Medical College, New York, New York
  - Montefiore-Einstein Cancer Center, The Bronx, New York
  - Levine Cancer Institute/Blumenthal Cancer Center, Charlotte, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Guthrie Clinic, Ltd., Sayre, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Santee Hematology Oncology, Inc., Sumter, South Carolina
  - Center for Biomedical Research, Knoxville, Tennessee
  - Sarah Cannon Research Institution, Nashville, Tennessee

REFERENCES:
- [Background] Yardley DA, Weaver R, Melisko ME, Saleh MN, Arena FP, Forero A, Cigler T, Stopeck A, Citrin D, Oliff I, Bechhold R, Loutfi R, Garcia AA, Cruickshank S, Crowley E, Green J, Hawthorne T, Yellin MJ, Davis TA, Vahdat LT. EMERGE: A Randomized Phase II Study of the Antibody-Drug Conjugate Glembatumumab Vedotin in Advanced Glycoprotein NMB-Expressing Breast Cancer. J Clin Oncol. 2015 May 10;33(14):1609-19. doi: 10.1200/JCO.2014.56.2959. Epub 2015 Apr 6. PMID 25847941